CLINICAL TRIAL: NCT04002804
Title: Phase I Clinical Trial Of Immunotherapy With Autologous Tumor Lysate-Loaded Dendritic Cells In Patients With Recurrence Of Glioblastoma Multiforme
Brief Title: Immunotherapy With Autologous Tumor Lysate-Loaded Dendritic Cells In Patients With Recurrence Of Glioblastoma Multiforme
Acronym: Dendr2
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Temozolomide does not favour immune response; secondary GBM to be excluded
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DENDR2
Record Dates: First submitted 2019-06-10; First posted 2019-07-01 (Actual); Last update posted 2019-07-01 (Actual); Status verified 2019-06

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Intervention Model Description: Phase I, 2-stage Simon design (Simon et al., 1997), single-centre, un-controlled, open label, non randomized study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Immunotherapy (Experimental): Autologous DC loaded with a autologous tumor lysate, in order to stimulate the immune response of the patient.
  Interventions: Biological: Dendritic Cells Vaccine

INTERVENTIONS:
Biological: Dendritic Cells Vaccine — Right after the surgical resection of the recurrent tumor, leukapheresis will be performed.
  At least 5x109 PBMC must be collected by leukapheresis, so as to make the whole immunotherapy schedule workable.
  Starting at week 3, immunotherapy will include 4 bi-weeekly vaccinations first (injections I, II, III, IV), two further monthly vaccinations (injections V, VI) and a final vaccination (injection VII) two months after the sixth one. Injections I, V, VI and VII will contain 10 million tumor lysate-loaded DC, while the others will be of 5 million cells only.
  Vaccine doses will be injected in the forearm of the patient.

SUMMARY:
Rationale of the Study: Treatment for GBM currently consists of surgical resection of the tumour mass followed by radio- and chemotherapy. Nonetheless overall prognosis still remains bleak, recurrence is universal, and recurrent GBM patients clearly need innovative therapies. Dendritic cells (DC) immunotherapy could represent a well-tolerated, long-term tumour-specific treatment to kill all (residual) tumour cells which infiltrate in the adjacent areas of the brain. Preclinical investigations for the development of therapeutic vaccines against high grade gliomas, based on the use of DC loaded with a mixture of glioma-derived tumor have been carried out in rat as well as in mouse models, showing the capacity to generate a glioma-specific immune response. Mature DC loaded with autologous tumor lysate have been used also for the treatment of patients with recurrent malignant brain tumors; no major adverse events have been registered.

Results about the use of immunotherapy for GBM patients are encouraging, but further studies are necessary to find out the most effective and safe combination of immunotherapy with radio- and chemotherapy after exeresis of the tumour mass.

Aim of the study: Primary objective of the study is to evaluate treatment tolerability and to get preliminary information about efficacy. Secondary objective is to evaluate the treatment effect on the immune response. Additional objective is to identify a possible correlation between methylation status of the MGMT promoter and tumor response to treatment.

A two-stage Simon design will be considered for the study. The primary objectives of the study include the evaluation of a PFS6 rate in treated patients. Assuming as outcome measure the percentage of PFS6 patients and of clinical interest an increase to 35% (P1) of the historical control response rate of 20% (P0), the null hypothesis will be rejected (a=0.05, b=0.2) at the end of the first stage if the response rate will be 5/22 treated patients (Fisher's exact test). In the second stage patients will be enrolled up to 72 overall. The study will be successful if at least 19 subjects out of 72 have PFS6 months after the beginning of the treatment.

DETAILED DESCRIPTION:
Study Design: Phase I, 2-stage Simon design (Simon et al., 1997), single-centre, un-controlled, open label, non randomized study.

The therapeutic program will include radical surgical resection of the tumor, followed by immunotherapy. Immunotherapy will comprise 4 biweekly vaccinations first (injections I, II, III, IV), 2 further monthly vaccinations (injections V, VI) and a final vaccination (injection VII) 2 months after the sixth one.

Injections I, V, VI and VII will contain 10 million tumor lysate-loaded DC, while the others will be of 5 million cells only. In correspondence to the third vaccine injection (week 7), 6 cycles of maintenance TMZ (mTMZ) will start. On the basis of the patient clinical status, further vaccine boosts will be considered as appropriate addition at the standard vaccination cycle.

Study Population: The first stage of the study will include 22 patients with recurrent GBM. The overall population at the end of the study will consist of 72 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders.
* Age 18 years and 70 years.
* Postoperative Karnofsky Performance Status >=70.
* Diagnosis of recurrent GBM (World Health Organization [WHO] grade IV astrocytoma).
* Diagnosis confirmed by the reference histopathology.
* Total or subtotal resection of tumor mass, confirmed by assessment of the neurosurgeon and by postoperative radiological assessment.
* Amount of non-necrotic tissue for lysate preparation and DC loading >= 1 gr, stored at -80°C.
* Corticosteroids daily dose <= 4 mg during the 2 days prior to leukapheresis.
* Life expectancy > 3 months.
* Signed informed consent.

Exclusion Criteria:

* Pregnancy.
* Participation in other clinical trials with experimental drugs simultaneously or within 1 month before this trial entry.
* Presence of acute infection requiring active treatment.
* Mandatory treatment with corticosteroids or salicylates in anti-inflammatory dose.
* Presence of sub-ependymal diffusion of the tumor.
* Haematology: leukocytes < 3,000/μl, lymphocytes < 500/μl, neutrophils < 1,000/μl, hemoglobin <9 g/100 ml, thrombocytes < 100,000/μl 2 days prior to leukapheresis.
* Documented immune deficiency.
* Documented autoimmune disease.
* Positive serology for HIV or hepatitis B or C.
* Allergies to any component of the DC vaccine.
* Known intolerance to TMZ.
* Other active malignancy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2010-04 (Actual); Primary Completion 2011-10 (Actual); Study Completion 2017-06-13 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Progression Free Survival at 6 Months (PFS-6) | Baseline to 6 months
  PFS-6 is defined as the percentage of participants with PFS at 6 months from the date of surgery for tumor recurrence to the first date of objectively determined progressive disease based on Response Assessment in Neuro-Oncology (RANO) criteria (Wen et al JCO 2010) or death from any cause. It is assumed that PFS follows an exponential distribution. Estimation using Kaplan-Meier analysis.

SECONDARY OUTCOMES:
Incidence of Treatment-related Adverse Events | Tolerability will be monitored throughout study completion, an average of 2 months
  Tolerability will be assessed using CTCAE version 3.0 and recording incidence, severity and type of adverse events.
Evaluation of the treatment effect on the immune response | Immune response will be monitored throughout study completion, an average of 2 months
  Levels of regulatory and CD8+ T cell in treated patients

IPD SHARING:
Plan to Share IPD: No